CLINICAL TRIAL: NCT02670005
Title: Fractional Flow Reserve Versus Angiography for Guiding Selective Percutaneous Coronary Intervention in ST-segment Elevation Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Jin Geng, MD, Nanjing Medical University
Other Study IDs: 20160010
Record Dates: First submitted 2016-01-26; First posted 2016-02-01 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-01

CONDITIONS: Fractional Flow Reserve; ST-segment Elevation Myocardial Infarction; Percutaneous Coronary Intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FFR-PCI group: patients with ST-segment elevation myocardial infarction (STEMI) who received fractional flow reserve (FFR)-guided selective percutaneous coronary intervention (PCI)
- angiography-PCI group: patients with STEMI who received angiography-guided selective PCI

SUMMARY:
To assess the outcomes of patients with ST-segment elevation myocardial infarction (STEMI) assigned to fractional flow reserve (FFR) and angiography-guided selective percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
The investigators retrospectively collect STEMI patients received selective PCI from Jan 2012 to Dec 2015. Clinical follow-up is performed from the date of FFR assessment to Dec 2016 or death, which is up to 5 years. The primary endpoint is major adverse cardiac events, composite of cardiac death, reinfarction and unplanned hospitalization due to cardiovascular reasons. The primary endpoints are cardiac death, reinfarction and unplanned hospitalization due to cardiovascular reasons. All deaths are considered cardiovascular unless an unequivocal noncardiac cause could be established. Reinfarction is defined as myocardial infarction after the PCI procedure. Unplanned hospitalization will be present only if the patient is hospitalized unexpectedly because of persisting or increasing complaints of angina, ventricular arrhythmias and heart failure. All patients were received FFR-guided PCI or angiography-guided PCI before enrollment, and the investigators do not assign specific interventions to the subjects during the study. So this study might be considered to be observational.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* documented acute ST-segment elevation myocardial infarction
* onset of symptom >6 days before percutaneous coronary intervention
* eligible for PCI

Exclusion Criteria:

* cardiogenic shock or hemodynamic instability
* highly tortuous or calcified arteries
* infarct related artery with a diameter < 2.5mm
* a life expectancy< 2 years
* intolerance to anti-platelet drugs
* left main disease (≥ 50% stenosis)
* contraindication to adenosine
* hypertrophic cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with ST-segment elevation myocardial infarction received selective percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | up to 5 years
  composite of cardiac death, reinfarction and unplanned hospitalization due to cardiovascular reasons

SECONDARY OUTCOMES:
cardiac death | up to 5 years
  All deaths are considered cardiovascular unless an unequivocal noncardiac cause could be established.
reinfarction | up to 5 years
  Reinfarction is defined as myocardial infarction after the PCI procedure.
unplanned hospitalization due to cardiovascular reasons | up to 5 years
  Unplanned hospitalization will be present only if the patient is hospitalized unexpectedly because of persisting or increasing complaints of angina, ventricular arrhythmias and heart failure.

IPD SHARING:
Plan to Share IPD: No